CLINICAL TRIAL: NCT00249951
Title: Alkaline Citrate Treatment to Lower the Risk of Nephrocalcinosis in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. B. Hoppe, Head, Division of Pediatric Nephrology, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FG03-157
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Nephrocalcinosis
Keywords: nephrocalcinosis; premature infants; hypocitraturia; alcaline citrate therapy; Nephrocalcinosis in premature infants
MeSH Terms: conditions — Nephrocalcinosis; Premature Birth | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alkaline citrate — Prophylactic alkaline citrate medication during the first 8 weeks of life versus placebo solution to prevent nephrocalcinosis of prematurity.
  Other Names: no brand names, Shol's solution versus placebo solution (NaCl 0.9 %)

SUMMARY:
Preterm infants are at risk to develop nephrocalcinosis. Incidence numbers vary according to birth weight and gestation age. Very low birth weight infants have the highest risk index, with ~ 7-10 % of preterm infants developing nephrocalcinosis in the patient population. We, the researchers at the University of Cologne, and others found significantly decreased urinary citrate excretion (hypocitraturia) to be one of the main risk factors. Hence, we hypothesized, that prophylactic treatment with oral alkaline citrate solution (Shol's solution) would help to 1) increase urinary citrate excretion and 2) help to decrease the incidence of nephrocalcinosis.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 32 weeks gestation age and < 1500 g birth weight

Exclusion Criteria:

* Cardial, renal or gastrointestinal malformations
* Chronic renal failure
* Therapy with vitamin B6
* High dose treatment with furosemide or dexamethasone
* Addison's disease
* Severe metabolic alkalosis
* Worse clinical condition of preterm infant, which makes oral feeding impossible
* Participation in other studies

Ages: 5 Days to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Prevention of nephrocalcinosis | First eight weeks of life
  Prevention of the development of nephrocalcinosis under prophylactic treatment with an alkaline citrate prepration.

SECONDARY OUTCOMES:
Increase in urinary citrate excretion | First eight weeks of life
  Increase in urinary citrate excretion under prophylactic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hoppe, Prof. Dr., Principal Investigator — University Children's Hospital Cologne, Kerpenerstr. 62, D-50924 Cologne, Germany
Locations (1):
- Prof. Dr. Bernd Hoppe, Cologne, Germany

REFERENCES:
- [Background] Sikora P, Roth B, Kribs A, Michalk DV, Hesse A, Hoppe B. Hypocitraturia is one of the major risk factors for nephrocalcinosis in very low birth weight (VLBW) infants. Kidney Int. 2003 Jun;63(6):2194-9. doi: 10.1046/j.1523-1755.2003.t01-4-00001.x. PMID 12753307
- [Background] Hoppe B, Duran I, Martin A, Kribs A, Benz-Bohm G, Michalk DV, Roth B. Nephrocalcinosis in preterm infants: a single center experience. Pediatr Nephrol. 2002 Apr;17(4):264-8. doi: 10.1007/s00467-001-0816-8. PMID 11956879
- [Background] Hoppe B, Roth B, Bauerfeld C, Langman CB. Oxalate, citrate, and sulfate concentration in human milk compared with formula preparations: influence on urinary anion excretion. J Pediatr Gastroenterol Nutr. 1998 Oct;27(4):383-6. doi: 10.1097/00005176-199810000-00002. PMID 9779963
- [Background] Hoppe B, Hesse A, Neuhaus T, Fanconi S, Forster I, Blau N, Leumann E. Urinary saturation and nephrocalcinosis in preterm infants: effect of parenteral nutrition. Arch Dis Child. 1993 Sep;69(3 Spec No):299-303. doi: 10.1136/adc.69.3_spec_no.299. PMID 8215570